CLINICAL TRIAL: NCT00520546
Title: Clinical Value of [18]Fluoroethylcholine Positron-Emission-Tomography Combined With Endorectal Magnetic Resonance Imaging by Software Fusion for Pre-therapeutic Staging of Prostate Cancer
Brief Title: Clinical Value of FEC-PET Combined With Endorectal MRI for Pre-therapeutic Staging of Prostate Cancer
Acronym: FEC-PET/MRI
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Dr. Markus Hartenbach (Other)
Responsible Party: Sponsor-Investigator, Dr. Markus Hartenbach, Major Medical Corps and assistant medical director of the nuclear medicine department, German Federal Armed Forces
Organization: German Federal Armed Forces (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 12K3-S-140708; 2006-003933-33 (EudraCT Number)
Record Dates: First submitted 2007-08-23; First posted 2007-08-24 (Estimated); Results first posted 2012-06-20 (Estimated); Last update posted 2012-06-20 (Estimated); Status verified 2012-06

CONDITIONS: Prostate Cancer
Keywords: PET; MRI; Choline; FEC; prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): Patients with prostate carcinoma confirmed by needle biopsy, age >50 years, planned radical prostatectomy with lymph-node dissection, fasting for >12 hours before FEC-PET and an interval between biopsy and PET >3 weeks.
  Interventions: Other: 18F-Ethylcholine Positron Emission Tomography (FEC-PET); Other: Endorectal Magnetic Resonance Imaging (1.5Tesla) (eMRI)

INTERVENTIONS:
Other: 18F-Ethylcholine Positron Emission Tomography (FEC-PET) — PET scans were performed on a LSO scanner (ECAT ACCEL, Siemens, Erlangen, Germany) by using a multiphase protocol starting with a "cold" transmission scan of the lower pelvis. This was followed by a list mode emission scan with 10 frames à 1 minute starting immediately after the administration of 3.3MBq [18F]Fluoroethylcholine chloride (FEC; Eckert & Ziegler EURO-PET Berlin GmbH) as a bolus through the cubital vein. After a short gap due to computer processing time the whole body scan was performed starting at the upper thoracic aperture down to the proximal femur. Acquisition parameters were 3 minutes emission scan and 2 minutes transmission scan for each bed position. Therefore the prostate region was scanned again at 45 minutes p.i. (post injection) A delayed local acquisition at 65 minutes over the lower pelvis with 6 minutes emission and 2 minutes transmission finished the diagnostic acquisition procedure.
Other: Endorectal Magnetic Resonance Imaging (1.5Tesla) (eMRI) — The MRI examination was performed on a 1.5Tesla MRI system (Gyroscan ACS-NT, Philips, Hamburg, Germany) with combined QBody and endorectal coil. Pelvic assessment and lymph node staging was effected with 5mm T2 weighted (T2w) turbo spin echo (TSE) transversal and a coronal short-tau inversion recovery (STIR) sequence. For prostate assessment, 3mm endorectal T2w spin echo (SE) sagittal, transversal and coronal sequences were acquired.

SUMMARY:
To investigate the sensitivity of the [18F]fluoroethylcholine (FEC) Positron-Emission-Tomography/ Magnetic Resonance Imaging (PET/MRI) method in tumour detection and location (side assignment, encapsulation, invasion of the seminal vesicle) and detection of affected lymph nodes, and to compare these with presently used detection procedures (needle biopsy, digital rectal examination, transrectal ultrasound, and pre-therapeutic assessment), with a view to finding out whether the [18F]fluoroethylcholine PET/MRI method is comparable to, or superior to, the established method. Postoperative histology served as the standard of reference.

DETAILED DESCRIPTION:
Prostate carcinoma is today in Germany the most frequently diagnosed cancer disease of men and is - after bronchial carcinoma - their second most frequent cause of cancer-related death. Around 22% of all new cancer diagnoses among males are prostate-related. This corresponds to an age-adjusted incidence rate of nearly 100 per 100,000 males in the population, and to well above 40,000 new diagnoses of prostate cancer per year [Robert-Koch-Institut, 2010]. The dramatic increase in recent decades is attributable more to improved diagnostic methods and a generally increased life expectancy than to an actual increase in the incidence of disease [Robert-Koch-Institut, 2010].

The total annual mortality rate is around 11,000 [Statistisches Bundesamt, 1994]. Prostate carcinoma is virtually unknown among men under 40 years of age. The annual prevalence rises with increasing age - between the 40th and 80th years of life by a factor of more than 1000. Autopsies have shown that among men over 70 up to 80% have a latent prostate carcinoma, without it being fatal [Breslow 1977; Börgemann, 2006]. The patients' average age at diagnosis is 71 years.

The five-year prostate-cancer-specific survival rate after diagnosis is about 80-99% for tumours that are restricted to the gland itself [Porter, 2006]. For disseminated tumours this figure is considerably smaller, not more than 35% [von Eschenbach, 1996]. A prospect of complete regression exists only for non-metastasing carcinomas, but there it is quite good: under aggressive treatment, 90% of cancers restricted to the prostate itself can be completely cured, as can 50% of those that have crossed the gland's capsule [Deutsche Gesellschaft für Urologie, 2009].

At present, there is a lack of adequate pre-therapeutic staging methods. This in turn often prevents the reliable choice of a stage-adapted therapeutic regimen, which could possibly offer a better prognosis even for carcinomas extending into neighbouring organs. A consequence of this uncertainty is that in individual cases the therapy is not ideally suited to the stage of disease, and the success of radiation treatment, hormonal therapy and chemotherapy can only approximately be matched with the stage of dissemination. Until now, the only reliable method for lymph-node diagnosis is operative staging by lymphadenectomy. No reliable diagnostic method is available by which the degree of spreading of the tumour within the prostate can be established.

In this context, Positron-Emission-Tomography (PET) examination with radioactively labelled choline appears to offer a promising primary imaging-diagnostic staging method, as indicated by the studies reviewed below. This diagnostic method as applied to humans was first described by Gauthier et al. [1985]. This was followed by two detailed reports from a Japanese group: Hara et al. [1997] first investigated the potential of [11C]choline in brain tumours and found a clear enrichment of this marker in the tumours of 24 patients, while normal brain tissue was not enriched with it. In a subsequent study by the same group [Hara, 1998], the enrichment of fluorodeoxyglucose was compared with the choline uptake in the lesions of ten prostate-cancer patients. Thus, the choline enrichment (SUV, standardised uptake value) was 3.48 ± 1.31 in 43 lesions, while in the normal environment of the lesser pelvis the corresponding value was below 1.0. De Jong et al. [2003] investigated 67 patients, of whom 15 had histologically confirmed lymph-node metastases: the [11C]choline test gave a 'true positive' result in 12 of 15 patients and a 'false negative' in 3 patients, thus indicating that [11C]choline PET is sufficiently sensitive and specific for the pre-operative staging of lymph-node metastases of prostate carcinoma. In a pre-operative staging using Magnetic Resonance Imaging (MRI) with a combined endorectal and body-phased-array coil, Pegios et al. [2003] investigated 42 patients with strong clinical suspicion, or with needle-biopsy confirmation, of prostate cancer and were able to differentiate between stages of extracapsular growth and seminal-vesicle infiltration (tumor stage T2 versus T3 [T2=tumor restricted to the gland itself; T3a=extracapsule growing of the tumor; T3b= tumor infiltration into the seminal-vesicles]) with an accuracy of 94-97% (sensitivity 100%, specificity between 87% and 93% for observers 1 and 2). The exact, local tumour stage was identified with an accuracy of 75%. However, for lymph-node infiltration a sensitivity of only 25% was achieved: one of four lymph-node-positive patients was correctly identified. In a more recent study, a Japanese group [Yamaguchi, 2005] investigated the application of nuclear magnetic resonance (NMR) spectroscopy, magnetic resonance imaging (MRI) and choline-PET in 20 patients with needle-biopsy-confirmed prostate cancer. The PET imaging achieved a sensitivity of 100%, NMR (quotient [(creatine + choline) / citrate]) 65% and unsupported MRI 60%. For 16 patients radical prostatectomy was performed; results correlated with those of pre-operative local staging with PET by 81%, and with MRI by 50%. The site of choline uptakes in PET was visualised by MRI using the distance of the prostate from the femoral head and the pubic symphysis.At present, no data relevant for the present study indication are available on the software-fused imaging by combined PET/MRI. The combination of high-resolution endorectal MRI with functional PET imaging could come to offer a decisive advantage in the staging of prostate carcinoma. The present study was designed to test this in an appropriate patient population.

A system combining PET and MRI was recently granted approval in the U.S.A. by the U.S. Food and Drug Administration [FDA, 2011].

ELIGIBILITY:
Inclusion Criteria:

* Histologically diagnosed prostate cancer (needle biopsy)
* Radical prostatectomy as primary treatment
* No nutrition within 12 hours before Positron-Emission-Tomography (PET)
* No food containing choline within 24 hous before PET
* Age > 50 years

Exclusion Criteria:

* Total endo-prothesis of the hip region
* Clinical or chemical detection of an acute infection
* Missing patient agreement
* Secondary cancer
* Surgical treatment within 3 month before PET
* Claustrophobia
* Medical drugs with choline
* Severe liver damage
* Cardiac infarction
* Bradycardia (pulse rate < 55/min)
* Allergic reaction against Neurotropan
* Bronchial asthma
* Cardiac pacemaker
* Small metal implants (e.g., clips, cochlea-implants, etc.)

Min Age: 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2007-12; Primary Completion 2011-02 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Markus Hartenbach, Dr., Principal Investigator — German Federal Armed Forces Hospital, Ulm, Dep. of Nuclear Medicine; Christoph Sparwasser, Prof. Dr., Study Director — German Federal Armed Forces Hospital Ulm, Dep. of Urology
Locations (1):
- German Federal Armed Forces Hospital, Ulm, Baden-Wurttemberg, Germany

REFERENCES:
- [Background] Robert-Koch-Institut (2010): Krebs in Deutschland 2005/2006 Häufigkeiten und Trends. A collaborative publication of the Robert-Koch-Institut and the Gesellschaft der epidemiologischen Krebsregister in Deutschland e.V. [Society for epidemiological cancer register], 7th edition, Berlin.
- [Background] Börgermann C, Rübben H (2006): Früherkennung des Prostatakarzinoms [Early recognition of prostate carcinoma]. Dtsch Arztebl. 103: 2399-2406.
- [Background] Breslow N, Chan CW, Dhom G, Drury RA, Franks LM, Gellei B, Lee YS, Lundberg S, Sparke B, Sternby NH, Tulinius H. Latent carcinoma of prostate at autopsy in seven areas. The International Agency for Research on Cancer, Lyons, France. Int J Cancer. 1977 Nov 15;20(5):680-8. doi: 10.1002/ijc.2910200506. PMID 924691
- [Background] de Jong IJ, Pruim J, Elsinga PH, Vaalburg W, Mensink HJ. Preoperative staging of pelvic lymph nodes in prostate cancer by 11C-choline PET. J Nucl Med. 2003 Mar;44(3):331-5. PMID 12620996
- [Background] Deutsche Gesellschaft für Urologie (2009): Interdisziplinäre Leitlinie der Qualität S3 zur Früherkennung, Diagnose und Therapie der verschiedenen Stadien des Prostatakarzinoms [Interdisciplinary guideline for the early recognition, diagnosis and therapy of the various stages of prostate carcinoma]. Deutsche Gesellschaft für Urologie e. V. (ed.), p. 53 ff.
- [Background] FDA (2011): FDA clears new system to perform simultaneous PET, MRI scans. Available on-line at http://www.fda.gov/NewsEvents/Newsroom/PressAnnouncements/2011/ucm258700.htm
- [Background] Gauthier S, Diksic M, Yamamoto L, Tyler J, Feindel WH (1985): Positron emission tomography with [11C]-choline in human subjects. Can J Neurol Sci 12: 214.
- [Background] Hara T, Kosaka N, Shinoura N, Kondo T. PET imaging of brain tumor with [methyl-11C]choline. J Nucl Med. 1997 Jun;38(6):842-7. PMID 9189127
- [Background] Hara T, Kosaka N, Kishi H. PET imaging of prostate cancer using carbon-11-choline. J Nucl Med. 1998 Jun;39(6):990-5. PMID 9627331
- [Background] Hara T, Kosaka N, Kishi H. Development of (18)F-fluoroethylcholine for cancer imaging with PET: synthesis, biochemistry, and prostate cancer imaging. J Nucl Med. 2002 Feb;43(2):187-99. PMID 11850483
- [Background] Kwee SA, Coel MN, Lim J, Ko JP. Prostate cancer localization with 18fluorine fluorocholine positron emission tomography. J Urol. 2005 Jan;173(1):252-5. doi: 10.1097/01.ju.0000142099.80156.85. PMID 15592091
- [Background] Pegios W, Bentas W, Wittmann L, Mack MG, Zangos S, Sollner O, Binder J, Fellbaum C, Jonas D, Vogl TJ. [MRI staging of prostate cancer with the combined endorectal body phased-array coil and histologic correlation]. Rofo. 2003 Dec;175(12):1660-6. doi: 10.1055/s-2003-45325. German. PMID 14661137
- [Background] Porter CR, Kodama K, Gibbons RP, Correa R Jr, Chun FK, Perrotte P, Karakiewicz PI. 25-year prostate cancer control and survival outcomes: a 40-year radical prostatectomy single institution series. J Urol. 2006 Aug;176(2):569-74. doi: 10.1016/j.juro.2006.03.094. PMID 16813891
- [Background] Yamaguchi T, Lee J, Uemura H, Sasaki T, Takahashi N, Oka T, Shizukuishi K, Endou H, Kubota Y, Inoue T. Prostate cancer: a comparative study of 11C-choline PET and MR imaging combined with proton MR spectroscopy. Eur J Nucl Med Mol Imaging. 2005 Jul;32(7):742-8. doi: 10.1007/s00259-004-1755-y. Epub 2005 Mar 15. PMID 16052370

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment of first patient: 18th. December, 2007 Completion by last patient: 12th. January, 2011 Single Center Study at Federal Armed Forces Hospital Ulm
Pre-assignment Details: 44 patients were enrolled, 38 patients completed the study. 1 patient decided not to choose prostatectomy after Positron-Emission-Tomography/ Magnetic Resonance Imaging (PET/MRI), although it was planned at point of enrollment. 5 patients did not get a PET/MRI-can because of failed radiopharmaceutical synthesis of [18F]fluoroethylcholine (FEC).
Groups:
- FEC-PET/eMRI: The day before surgery, fasting patients received a bladder catheter right before Positron-Emission-Tomography/ Magnetic Resonance Imaging (PET/MRI) examination to avoid different sizes of the urinary bladder in PET and MRI scan and to reduce bladder FEC-activity overlay of the prostate. After applying the endorectal MRI coil patients were positioned in a vacuum mattress on MRI table. Additionally, 4 PET/MRI multimodality spot markers containing 37kBq [22Na] and a MRI T2w (T2 weighed) hyperintense gel were attached at the hip region to allow landmark PET/MRI fusion. After MRI acquisition the modular MRI table was fixed on the PET table system. Patients kept in the same position during the whole procedure. PET scans were performed by using a multiphase protocol starting with a list mode emission scan immediately after the administration of 3.3MBq [18F]fluoroethylcholine (FEC) as a bolus through the cubital vein.
Period: Overall Study
Arm/Group | FEC-PET/eMRI
Started | 44
Completed | 38
Not Completed | 6
Not completed — Withdrawal by Subject | 1
Not completed — failed radiopharmaceut. synthesis of FEC | 5

BASELINE CHARACTERISTICS:
Arm/Group | FEC-PET/eMRI
Number analyzed (Participants) | 44
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 23
  >=65 years | 21
Age Continuous [Mean (Standard Deviation); unit: years] | 65 (6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 44
Region of Enrollment [Number; unit: participants]
  Germany | 44

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Positive or Negative Results in PET, MRI or PET/MRI for Prostate Cancer Compared to Histological Findings
Description: PET positive lesions were measured on its own and evaluated as malignant just as hypointense lesions on MRI. In PET/MRI analysis, MRI suspect lesions without FEC uptake were considered not to be malignant. PET positive lesions in central periurethral zone with inhomogenous signal intensity and sharp edges on MRI images were also considered to be benign. PET positive lesions in the peripheral zone without a hypointense correlate on MRI were considered to be malignant. At least 1 histological confirmed cancer lesion has to be detected by each of the 3 methods to be patient based true positive.
Time Frame: within < 2 weeks after PET/MRI
Population: Comparison of imaging results (FEC-PET, MRI and PET/MRI) with postoperative histological findings (all patients).
Measure: Number; unit: participants
Groups:
- [18F]Fluoroethylcholine Positron-Emission-Tomography (FEC-PET): PET scans were performed on a LSO scanner (ECAT ACCEL, Siemens, Erlangen, Germany) by using a multiphase protocol starting with a "cold" transmission scan of the lower pelvis. This was followed by a list mode emission scan with 10 frames à 1 minute starting immediately after the administration of 3.3MBq [18F]Fluoroethylcholine chloride (FEC; Eckert & Ziegler EURO-PET Berlin GmbH) as a bolus through the cubital vein. Acquisition parameters were 3 minutes emission scan and 2 minutes transmission scan for each bed position. Therefore the prostate region was scanned again at 45 minutes p.i. (post injection) A delayed local acquisition at 65 minutes over the lower pelvis with 6 minutes emission and 2 minutes transmission finished the diagnostic acquisition procedure.
- Magnetic Resonance Imaging (MRI): The MRI examination was performed on a 1.5Tesla MRI system (Gyroscan ACS-NT, Philips, Hamburg, Germany) with combined QBody and endorectal coil. Pelvic assessment and lymph node staging was effected with 5mm T2 weighted (T2w) turbo spin echo (TSE) transversal and a coronal short-tau inversion recovery (STIR) sequence. For prostate assessment, 3mm endorectal T2 weighed (T2w) spin echo (SE) sagittal, transversal and coronal sequences were acquired. Transversal sequences were angulated 90° to intraprostatic bladder catheter to allow exact correlation with histological holoptical slices.
- PositronEmissionTomography/MagneticResonanceImaging (PET/MRI): PET images at 45 min p.i. (post injection) and 65 min p.i. were fused with transversal endorectal and QBody T2 weighed (T2w) MRI images by using Hermes Medical Solutions Multi Modality landmark fusion tool. The four PET/MRI spot markers served as references. Without any patient movement between both modalities the fused images fitted exactly.
Arm/Group | [18F]Fluoroethylcholine Positron-Emission-Tomography (FEC-PET) | Magnetic Resonance Imaging (MRI) | PositronEmissionTomography/MagneticResonanceImaging (PET/MRI)
Number analyzed (Participants) | 38 | 38 | 38
participants
  True Positive | 36 | 26 | 35
  False Positive | 1 | 1 | 0
  True Negative | 0 | 0 | 1
  False Negative | 1 | 11 | 2
  Total True | 36 | 27 | 36
  Total False | 2 | 11 | 2
Statistical Analysis 1: Comparison: [18F]Fluoroethylcholine Positron-Emission-Tomography (FEC-PET); results from FEC-PET as compared with histological results on a patient based analysis Null hypothesis: patient distribution in contingency table is incidental; Test type: Superiority or Other; p = 0.0526, Fisher Exact; sensitivity = 97, 95% CI 2-sided [86 to 100]
Statistical Analysis 2: Comparison: [18F]Fluoroethylcholine Positron-Emission-Tomography (FEC-PET); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0526, Fisher Exact; specificity = 0, 95% CI 2-sided [0 to 98]
Statistical Analysis 3: Comparison: [18F]Fluoroethylcholine Positron-Emission-Tomography (FEC-PET); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0526, Fisher Exact; accuracy = 95, 95% CI 2-sided [82 to 99]
Statistical Analysis 4: Comparison: Magnetic Resonance Imaging (MRI); results from MRI as compared with histological results on a patient based analysis Null hypothesis: patient distribution in contingency table is incidental; Test type: Superiority or Other; p < 0.0001, Fisher Exact; sensitivity = 70, 95% CI 2-sided [53 to 84]
Statistical Analysis 5: Comparison: Magnetic Resonance Imaging (MRI); [analysis description as in outcome 1, analysis 4]; Test type: Superiority or Other; p < 0.0001, Fisher Exact; specificity = 0, 95% CI 2-sided [0 to 98]
Statistical Analysis 6: Comparison: Magnetic Resonance Imaging (MRI); [analysis description as in outcome 1, analysis 4]; Test type: Superiority or Other; p < 0.0001, Fisher Exact; accuracy = 68, 95% CI 2-sided [51 to 83]
Statistical Analysis 7: Comparison: PositronEmissionTomography/MagneticResonanceImaging (PET/MRI); results from PET/MRI as compared with histological results on a patient based analysis Null hypothesis: patient distribution in contingency table is incidental; Test type: Superiority or Other; p = 0.0043, Fisher Exact; sensitivity = 95, 95% CI 2-sided [82 to 99]
Statistical Analysis 8: Comparison: PositronEmissionTomography/MagneticResonanceImaging (PET/MRI); [analysis description as in outcome 1, analysis 7]; Test type: Superiority or Other; p = 0.0043, Fisher Exact; specificity = 100, 95% CI 2-sided [3 to 100]
Statistical Analysis 9: Comparison: PositronEmissionTomography/MagneticResonanceImaging (PET/MRI); [analysis description as in outcome 1, analysis 7]; Test type: Superiority or Other; p = 0.0043, Fisher Exact; accuracy = 95, 95% CI 2-sided [82 to 99]

2. Secondary Outcome: Lesion Based Analysis of FEC-PET, Endorectal MRI and Combined FEC-PET/eMRI in All Patients
Description: PET positive lesions (n=128) were measured on its own and evaluated as malignant just as hypointense lesions on MRI. In PET/MRI analysis, MRI suspect lesions without FEC uptake were considered not to be malignant. PET positive lesions in central periurethral zone with inhomogenous signal intensity and sharp edges on MRI images were also considered to be benign. PET positive lesions in the peripheral zone without a hypointense correlate on MRI were considered to be malignant. Sensitivity, specificity, accuracy, negative and positive predictive values were determined.
Time Frame: within < 2 weeks after PET/MRI
Population: Comparison of lesion based (128)imaging results (FEC-PET, MRI and PET/MRI) with postoperative histological findings (all patients = 38).
Measure: Number; unit: lesions
Units Other Than Participants: lesions
Groups:
- FEC-PET: PET scans were performed on a LSO scanner (ECAT ACCEL, Siemens, Erlangen, Germany) by using a multiphase protocol starting with a "cold" transmission scan of the lower pelvis. This was followed by a list mode emission scan with 10 frames à 1 minute starting immediately after the administration of 3.3MBq [18F]Fluoroethylcholine chloride (FEC; Eckert & Ziegler EURO-PET Berlin GmbH) as a bolus through the cubital vein. Acquisition parameters were 3 minutes emission scan and 2 minutes transmission scan for each bed position. Therefore the prostate region was scanned again at 45 minutes p.i. (post injection) A delayed local acquisition at 65 minutes over the lower pelvis with 6 minutes emission and 2 minutes transmission finished the diagnostic acquisition procedure.
- Magnetic Resonance Imaging (MRI): The MRI examination was performed on a 1.5Tesla MRI system (Gyroscan ACS-NT, Philips, Hamburg, Germany) with combined QBody and endorectal coil. Pelvic assessment and lymph node staging was effected with 5mm T2w TSE transversal and a coronal STIR sequence. For prostate assessment, 3mm endorectal T2w SE sagittal, transversal and coronal sequences were acquired. Transversal sequences were angulated 90° to intraprostatic bladder catheter to allow exact correlation with histological holoptical slices.
- PET/MRI: PET images at 45 min p.i. and 65 min p.i. (post injection) were fused with transversal endorectal and QBody T2w MRI images by using Hermes Medical Solutions Multi Modality landmark fusion tool. The four PET/MRI spot markers served as references. Without any patient movement between both modalities the fused images fitted exactly.
Arm/Group | FEC-PET | Magnetic Resonance Imaging (MRI) | PET/MRI
Number analyzed (Participants) | 38 | 38 | 38
Number analyzed (lesions) | 128 | 128 | 128
lesions
  True positive | 59 | 40 | 55
  False positive | 26 | 27 | 8
  True negative | 19 | 18 | 37
  False negative | 24 | 43 | 28
  Total true | 78 | 58 | 92
  Total false | 50 | 70 | 36
Statistical Analysis 1: Comparison: FEC-PET; lesion based (all lesions = 128) results from FEC-PET as compared with histological results on a lesion based analysis of all patients (38) Null hypothesis: patient distribution in contingency table is incidental; Test type: Superiority or Other; p = 0.09, Fisher Exact; positive prediction = 69
Statistical Analysis 2: Comparison: FEC-PET; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.09, Fisher Exact; negative prediction = 44
Statistical Analysis 3: Comparison: FEC-PET; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.09, Fisher Exact; sensitivity = 71
Statistical Analysis 4: Comparison: FEC-PET; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.09, Fisher Exact; specificity = 42
Statistical Analysis 5: Comparison: FEC-PET; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.09, Fisher Exact; accuracy = 61
Statistical Analysis 6: Comparison: Magnetic Resonance Imaging (MRI); lesion based (all lesions = 128) results from MRI as compared with histological results on a lesion based analysis of all patients (38) Null hypothesis: patient distribution in contingency table is incidental; Test type: Superiority or Other; p = 0.27, Fisher Exact; positive prediction = 60
Statistical Analysis 7: Comparison: Magnetic Resonance Imaging (MRI); [analysis description as in outcome 2, analysis 6]; Test type: Superiority or Other; p = 0.27, Fisher Exact; negative prediction = 30
Statistical Analysis 8: Comparison: Magnetic Resonance Imaging (MRI); [analysis description as in outcome 2, analysis 6]; Test type: Superiority or Other; p = 0.27, Fisher Exact; sensitivity = 48
Statistical Analysis 9: Comparison: Magnetic Resonance Imaging (MRI); [analysis description as in outcome 2, analysis 6]; Test type: Superiority or Other; p = 0.27, Fisher Exact; specificity = 40
Statistical Analysis 10: Comparison: Magnetic Resonance Imaging (MRI); [analysis description as in outcome 2, analysis 6]; Test type: Superiority or Other; p = 0.27, Fisher Exact; accuracy = 45
Statistical Analysis 11: Comparison: PET/MRI; lesion based (all lesions = 128) results from PET/MRI as compared with histological results on a lesion based analysis of all patients (38) Null hypothesis: patient distribution in contingency table is incidental; Test type: Superiority or Other; p < 0.001, Fisher Exact; positive prediction = 87
Statistical Analysis 12: Comparison: PET/MRI; [analysis description as in outcome 2, analysis 11]; Test type: Superiority or Other; p < 0.001, Fisher Exact; negative prediction = 57
Statistical Analysis 13: Comparison: PET/MRI; [analysis description as in outcome 2, analysis 11]; Test type: Superiority or Other; p < 0.001, Fisher Exact; sensitivity = 66
Statistical Analysis 14: Comparison: PET/MRI; [analysis description as in outcome 2, analysis 11]; Test type: Superiority or Other; p < 0.001, Fisher Exact; specificity = 82
Statistical Analysis 15: Comparison: PET/MRI; [analysis description as in outcome 2, analysis 11]; Test type: Superiority or Other; p < 0.001, Fisher Exact; accuracy = 72

3. Secondary Outcome: Lesion Based Analysis of FEC-PET, Endorectal MRI and Combined FEC-PET/eMRI in Patients With Gleason Score >6 (3+3)
Description: PET positive lesions in patients with Gleason >6(3+3),n=43 were measured on its own and evaluated as malignant just as hypointense lesions on MRI. In PET/MRI analysis, MRI suspect lesions without FEC uptake were considered not to be malignant. PET positive lesions in central periurethral zone with inhomogenous signal intensity and sharp edges on MRI images were also considered to be benign. PET positive lesions in the peripheral zone without a hypointense correlate on MRI were considered to be malignant. Sensitivity, specificity, accuracy, negative & positive predictive values were determined.
Time Frame: within < 2 weeks after PET/MRI
Population: lesion based (patients with Gleasons Score >6(3+3),n= 43) results from FEC-PET as compared with histological results on a lesion based analysis of all patients (38).
  Gleason Grades: 1+2=well differentiated (rare), 3=moderately diff., 4=poorly diff., 5=undifferentiated
  Gleason Score = histological primary grade + secondary grade (min=2,max=10)
Measure: Number; unit: lesions
Units Other Than Participants: lesions
Arm/Group | FEC-PET | Magnetic Resonance Imaging (MRI) | PET/MRI
Number analyzed (Participants) | 38 | 38 | 38
Number analyzed (lesions) | 43 | 43 | 43
lesions
  True positive | 27 | 22 | 27
  False positive | 5 | 9 | 1
  True negative | 8 | 4 | 11
  False negative | 3 | 8 | 4
  Total true | 35 | 26 | 38
  Total false | 8 | 17 | 5
Statistical Analysis 1: Comparison: FEC-PET; Lesion based analysis of FEC-PET, endorectal MRI and combined FEC-PET/eMRI in patients with Gleason Score >6 (n=43) as compared with histological results on a lesion based analysis of all patients (38) Null hypothesis: patient distribution in contingency table is incidental; Test type: Superiority or Other; p < 0.001, Fisher Exact; positive prediction = 84
Statistical Analysis 2: Comparison: FEC-PET; Lesion based analysis of FEC-PET, endorectal MRI and combined FEC-PET/eMRI in patients with Gleason Score >6 (n=43) as compared with histological results on a lesion based analysis of all patients (n=38) Null hypothesis: patient distribution in contingency table is incidental; Test type: Superiority or Other; p < 0.001, Fisher Exact; negative prediction = 73
Statistical Analysis 3: Comparison: FEC-PET; [analysis description as in outcome 3, analysis 2]; Test type: Superiority or Other; p < 0.001, Fisher Exact; sensitivity = 90
Statistical Analysis 4: Comparison: FEC-PET; [analysis description as in outcome 3, analysis 2]; Test type: Superiority or Other; p < 0.001, Fisher Exact; specificity = 84
Statistical Analysis 5: Comparison: FEC-PET; [analysis description as in outcome 3, analysis 2]; Test type: Superiority or Other; p < 0.001, Fisher Exact; accuracy = 82
Statistical Analysis 6: Comparison: Magnetic Resonance Imaging (MRI); [analysis description as in outcome 3, analysis 2]; Test type: Superiority or Other; p = 0.53, Fisher Exact; positive prediction = 71
Statistical Analysis 7: Comparison: Magnetic Resonance Imaging (MRI); [analysis description as in outcome 3, analysis 2]; Test type: Superiority or Other; p = 0.53, Fisher Exact; negative prediction = 33
Statistical Analysis 8: Comparison: Magnetic Resonance Imaging (MRI); [analysis description as in outcome 3, analysis 2]; Test type: Superiority or Other; p = 0.53, Fisher Exact; sensitivity = 73
Statistical Analysis 9: Comparison: Magnetic Resonance Imaging (MRI); [analysis description as in outcome 3, analysis 2]; Test type: Superiority or Other; p = 0.53, Fisher Exact; specificity = 31
Statistical Analysis 10: Comparison: Magnetic Resonance Imaging (MRI); [analysis description as in outcome 3, analysis 2]; Test type: Superiority or Other; p = 0.53, Fisher Exact; accuracy = 60
Statistical Analysis 11: Comparison: PET/MRI; [analysis description as in outcome 3, analysis 2]; Test type: Superiority or Other; p < 0.001, Fisher Exact; positive prediction = 96
Statistical Analysis 12: Comparison: PET/MRI; [analysis description as in outcome 3, analysis 2]; Test type: Superiority or Other; p < 0.001, Fisher Exact; negative prediction = 73
Statistical Analysis 13: Comparison: PET/MRI; [analysis description as in outcome 3, analysis 2]; Test type: Superiority or Other; p < 0.001, Fisher Exact; sensitivity = 87
Statistical Analysis 14: Comparison: PET/MRI; [analysis description as in outcome 3, analysis 2]; Test type: Superiority or Other; p < 0.001, Fisher Exact; specificity = 92
Statistical Analysis 15: Comparison: PET/MRI; [analysis description as in outcome 3, analysis 2]; Test type: Superiority or Other; p < 0.001, Fisher Exact; accuracy = 88

4. Secondary Outcome: Lesion Based Analysis of FEC-PET, Endorectal MRI and Combined FEC-PET/eMRI in Patients With Malignant Lesions >5mm (n=98)
Description: PET positive lesions were measured on its own and evaluated as malignant just as hypointense lesions on MRI. In PET/MRI analysis, MRI suspect lesions without FEC uptake were considered not to be malignant. PET positive lesions in central periurethral zone with inhomogenous signal intensity and sharp edges on MRI images were also considered to be benign. PET positive lesions in the peripheral zone without a hypointense correlate on MRI were considered to be malignant. Sensitivity, specificity, accuracy, negative and positive predictive values were determined without malign lesions <=5mm.
Time Frame: within < 2 weeks after PET/MRI
Population: lesion based (malignant lesions >5mm, n=98) results from FEC-PET as compared with histological results on a lesion based analysis of all patients (38)
Measure: Number; unit: lesions
Units Other Than Participants: lesions
Arm/Group | FEC-PET | Magnetic Resonance Imaging (MRI) | PET/MRI
Number analyzed (Participants) | 38 | 38 | 38
Number analyzed (lesions) | 98 | 98 | 98
lesions
  True positive | 48 | 37 | 48
  False positive | 24 | 26 | 8
  True negative | 18 | 16 | 32
  False negative | 8 | 19 | 10
  Total true | 66 | 53 | 80
  Total false | 32 | 45 | 18
Statistical Analysis 1: Comparison: FEC-PET; Lesion based analysis of FEC-PET, endorectal MRI and combined FEC-PET/eMRI in patients with malign lesions >5mm (n=98) as compared with histological results on a lesion based analysis of all patients (n=38) Null hypothesis: patient distribution in contingency table is incidental; Test type: Superiority or Other; p = 0.002, Fisher Exact; positive prediction = 67
Statistical Analysis 2: Comparison: FEC-PET; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.002, Fisher Exact; negative prediction = 69
Statistical Analysis 3: Comparison: FEC-PET; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.002, Fisher Exact; sensitivity = 86
Statistical Analysis 4: Comparison: FEC-PET; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.002, Fisher Exact; specificity = 43
Statistical Analysis 5: Comparison: FEC-PET; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.002, Fisher Exact; accuracy = 67
Statistical Analysis 6: Comparison: Magnetic Resonance Imaging (MRI); [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.41, Fisher Exact; positive prediction = 59
Statistical Analysis 7: Comparison: Magnetic Resonance Imaging (MRI); [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.41, Fisher Exact; negative prediction = 46
Statistical Analysis 8: Comparison: Magnetic Resonance Imaging (MRI); [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.41, Fisher Exact; sensitivity = 66
Statistical Analysis 9: Comparison: Magnetic Resonance Imaging (MRI); [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.41, Fisher Exact; specificity = 38
Statistical Analysis 10: Comparison: Magnetic Resonance Imaging (MRI); [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.41, Fisher Exact; accuracy = 54
Statistical Analysis 11: Comparison: PET/MRI; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.001, Fisher Exact; positive prediction = 86
Statistical Analysis 12: Comparison: PET/MRI; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.001, Fisher Exact; negative prediction = 76
Statistical Analysis 13: Comparison: PET/MRI; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.001, Fisher Exact; sensitivity = 83
Statistical Analysis 14: Comparison: PET/MRI; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.001, Fisher Exact; specificity = 80
Statistical Analysis 15: Comparison: PET/MRI; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.001, Fisher Exact; accuracy = 82

ADVERSE EVENTS:
Time Frame: Enrollment of first patient: 18th. December, 2007 (before PET/MRI) Completion by last patient: 12th. January, 2011 (after surgery) During the whole period (3 years, 1 month) adverse event data were collected.
Arm/Group | FEC-PET/eMRI
Serious Adverse Events (participants affected / at risk) | 0/39
Other Adverse Events (participants affected / at risk) | 0/39

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No